CLINICAL TRIAL: NCT00962650
Title: A Feasibility Trial to Evaluate Natural Orifice Transgastric Endoscopic Diagnostic Peritoneoscopy With Laparoscopic Assistance.
Brief Title: Natural Orifice Transgastric Endoscopic (NOTES) Transgastric Diagnostic Peritoneoscopy With Laparoscopic Assistance
Acronym: NOTES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ethicon Endo-Surgery (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CI-08-0007
Record Dates: First submitted 2009-08-12; First posted 2009-08-20 (Estimated); Results first posted 2012-03-29 (Estimated); Last update posted 2012-03-29 (Estimated); Status verified 2012-03

CONDITIONS: Abdominal Adhesions
Keywords: abdominal adhesions; diagnostic peritoneoscopy; Natural Orifice Transluminal Endoscopic Surgery; NOTES

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- NOTES Toolbox (Experimental): Multiple devices designed for trans-orifice use during surgical procedures; used for transvaginal cholecystectomy in this trial
  Interventions: Device: Transgastric diagnostic peritoneoscopy with laparoscopic assistance

INTERVENTIONS:
Device: Transgastric diagnostic peritoneoscopy with laparoscopic assistance — Device: Natural Orifice Transgastric Endoscopic (NOTES GEN 1 Toolbox): Articulating Hook Knife(IN2505), Articulating Snare (IN2503), Articulating Needle Knife(IN2504), Articulating Graspers(IN2501 or IN2506), Articulating Biopsy Forceps(IN2502), Steerable Flexible Trocar (IN0501) with Rotary Access Needle (IN0502), Flexible Bipolar Hemostasis Forceps (IN0301), and/or Flexible Maryland Dissector(IN1601)

SUMMARY:
The study will document being able to successfully perform transgastric diagnostic peritoneoscopy (laparoscopic visualization) using a small collection of study surgical tools.

ELIGIBILITY:
Inclusion Criteria:

Men and women will be enrolled in this study who:

* Are willing to give consent and comply with evaluation and treatment schedule;
* At least 18 years of age;
* Are a candidate for surgical weight loss intervention (i.e. meet ASMBS and NIH criteria) for an RYGB procedure at the Investigational site;
* Have a history of open abdominal surgery or laparoscopic abdominal surgery;
* ASA Classification I, II, or III (Appendix II); and
* Have a negative serum pregnancy test (for women of childbearing potential).

Exclusion Criteria:

Subjects will be excluded from the study for any of the following:

* Use of immunosuppressive medications (within 6 months of surgery; single burst dosages and inhalable steroids are acceptable);
* Acute cholecystitis or acute pancreatitis;
* Evidence of abdominal abscess or mass;
* Diffuse peritonitis;
* Use of anticoagulants or anti-platelet agents (use of daily cardio protective doses of aspirin, up to 81 mg/day, is acceptable and shall not constitute an exclusion criterion) or the presence of coagulopathy;
* Clinical diagnosis of sepsis;
* Co-morbid condition(s) that could limit the subject's ability to participate in the study or to comply with follow-up requirements, or that could impact the scientific integrity of the trial;
* Planned concurrent surgical procedure other than RYGB or adhesiolysis;
* Prior or planned major surgical procedure within 30 days before or after study procedure;
* Participation in any other investigational device or drug trial that has not completed the primary endpoint or that clinically interferes with the current study endpoints;
* Previously enrolled in the current series of 4 trials investigating the EES NOTES GEN1 Toolbox; or
* Any condition which precludes compliance with the study (Investigator discretion).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2009-06; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey W Hazey, MD, FACS, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Medical Center, Columbus, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study Initiation Date: 09 June 2009 (First Informed consent signed) Study Completion Date:03 May 2010 (Last subject last visit) Enrollment Location: The Ohio State University Medical Center
Pre-assignment Details: All enrolled subjects provided informed consent to participate in the study, met protocol entry criteria, and had the study procedure attempted (ITT population).
Groups:
- Natural Orifice Transgastric Diagnostic Peritineoscopy: Natural orifice transgastric diagnostic peritineoscopy refers to performing diagnostic peritineoscopy with laparoscopic assistance with access through the stomach instead of using a trocar placed through the skin.
Period: Overall Study
Arm/Group | Natural Orifice Transgastric Diagnostic Peritineoscopy
Started | 10
Completed | 8
Not Completed | 2
Not completed — Transgastric DP was not completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Natural Orifice Transgastric Diagnostic Peritineoscopy
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 1
Age Continuous [Mean (Standard Deviation); unit: years] | 54.2 (9.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Completion of Diagnostic Peritineoscopy
Description: Number of participants in which transgastric access was achieved using the EES NOTES GEN1 Toolbox
  Outcome description: Completion of diagnostic peritoneoscopy after transgastric access was completed using a flexible, steerable trocar. Because this was a feasibility trial, transgastric access was the primary outcome.
Time Frame: Assessed intra-operatively as the time from first insertion of the flexible trocar into the oral cavity to final withdrawal of the flexible trocar
Population: The subject pool was limited to individuals scheduled for Rouen Y gastric bypass(Intent to Treat population). There was no statistical analysis. Success was based on completion of the diagnostic peritineoscopy procedure after transgastric access.
Measure: Number; unit: Participants
Arm/Group | Natural Orifice Transgastric Diagnostic Peritineoscopy
Number analyzed (Participants) | 10
Participants | 8

ADVERSE EVENTS:
Time Frame: Adverse events were collected from Study Initiation Date (first Informed Consent signed) 09 June 2009 until Study Completion Date (last participant's last visit) on 03 May 2010.
Arm/Group | Natural Orifice Transgastric Diagnostic Peritineoscopy
Serious Adverse Events (participants affected / at risk) | 1/10
Other Adverse Events (participants affected / at risk) | 0/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Natural Orifice Transgastric Diagnostic Peritineoscopy (N=10)
ESOPHAGEAL INJURY/ OESOPHAGEAL INJURY (Surgical and medical procedures) | 1 (1) — ESOPHAGEAL INJURY/ OESOPHAGEAL INJURY occurred when passing study device down esophagus.

LIMITATIONS AND CAVEATS:
Ten male and female subjects indicated for Diagnostic Peritoneoscopy in advance of Roux-en Y Gastic Bypass procedure, who had a history of previous abdominal surgery, and met study Inclusion Criteria, were enrolled in the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No